CLINICAL TRIAL: NCT06234540
Title: Effect of Autologous Platelet Rich Plasma(a-PRP) Intrauterine Instillation in Infertile Women With Thin Endometrium in Frozen-thawed Embryo Transfer Cycle: a Randomized Controlled Study
Brief Title: a-PRP Intrauterine Instillation in Women With Thin Endometrium
Acronym: PRP(a-PRP)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Sootthinan Pothisan, Infertility unit, Obstetric and gynecology department of Siriraj hospital, Mahidol university, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 853/2566(IRB4); WHO (Other: U1111-1303-0085)
Record Dates: First submitted 2024-01-23; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Thin Endometrium
Keywords: PRP, Platelet-rich plasma, IVF/ICSI, Frozen Thaw cycle

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- aPRP 1 (Experimental): a-PRP intrauterine instillation on Menstruation Cycle Day 8 during frozen thaw cycle procedure
  Interventions: Procedure: PRP
- aPRP 2 (Experimental): a-PRP intrauterine instillation on Menstruation Cycle Day 8 and Day 10 during frozen thaw cycle procedure
  Interventions: Procedure: PRP
- Controlled (Experimental): Standard treatment of frozen thaw cycle
  Interventions: Other: Standard treatment

INTERVENTIONS:
Procedure: PRP — a-PRP intrauterine instillation before frozen-thawed embryo transfer cycle
  Arms: aPRP 1; aPRP 2
Other: Standard treatment — Standard treatment
  Arms: Controlled

SUMMARY:
This study sought to compare the endometrial thickness among infertile women with a history of thin endometrium together with previous cancellation from IVF/ICSI inspection of intrauterine instillation of autologous-PRP or no treatment before embryo transfer in the frozen-thaw cycles.

DETAILED DESCRIPTION:
At present, infertility is a major problem in Thailand. As a result, the Ministry of Public Health has to push the guidelines for using reproductive technology to play a role in increasing the population in the country. The most well-known use of reproductive technology is In vitro fertilization (IVF) has a success rate of approximately 35-40%. There are many factors affecting the success of pregnancy, one of which is the thickness of the uterine cavity.

An endometrial thickness of less than 7 mm in the middle of the menstrual cycle is called endometrial lining. Thin endometrium, which can affect pregnancy Both the rate of embryo implantation pregnancy rate and miscarriage rates In the process of IVF In practice, the appropriate and popular thickness of the uterine cavity for embryo transfer is based on a thickness greater than equal to 7 mm. This is because many studies have found that the thickness of the uterine cavity At 8 mm, this can significantly increase pregnancy rates.

Platelet Rich Plasma (PRP) is another new treatment approach. There is information and research results that show that PRP can increase the thickness of the uterine cavity. and found to help increase blood flowing to the area The uterine wall in infertile women who have a thin uterine cavity. According to a study by Chang et al., in 2015, PRP was used to increase the thickness of the uterine cavity. Found that it can increase the thickness of the uterine cavity. It also tends to increase the pregnancy rate. This is likely caused by Helping increase the number of cells cell regeneration and repair of worn out parts of body cells Through the main mechanism of PRP is adding substances that stimulate cell growth (Growth factors) and proteins that are signals between cells (Cytokines). Someone has studied and compared the levels of substances that stimulate cell growth in PRP. Compared with lymph (plasma), it was found that the levels of cell growth stimulants in PRP were 2.4-2.8 times higher than those in lymph, with statistical significance.

Moreover, the process of preparing PRP is not complicated and the prepared ingredients do not cause any harmful side effects to the body. Therefore, it can be seen from various sectors and various studies that PRP has been used to accelerate growth, such as treating hair loss or baldness. Reducing inflammation or pain in various joints Or even use it to restore beauty, nourish the skin, etc.

In this study The authors therefore attempt to demonstrate the benefits of PRP that may promote endometrial thickening in women with endometrial hyperplasia in order to achieve appropriate endometrial thickness. Received embryo transfer in the next embryo freezing cycle. In addition, in Thailand there has never been a study of increasing the thickness of the uterine cavity with PRP injections before. Therefore, the creators expect that this method may be a method that can increase the implantation rate. Embryo or clinical pregnancy rate Including reducing the rate of embryo implantation cancellations to reduce anxiety for infertile couples in Thailand.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo frozen embryo transfer (Frozen-thawed cycle)
* Age above 18 years
* Thai nationality
* Have a history of cycle cancellation due to a thin endometrium <7 mm. after standard hormonal treatmetn

Exclusion Criteria:

* medical conditions eg. Platelet dysfunction , vWD
* thrombocytopenia <100,000 cell/mm3
* Receive antiplatelet therapy
* Uterine anomaly, cavity distortion eg submucous myoma uteri, uterine synergia, endometrial polyp

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — infertile woman
Enrollment: 36 (Estimated)
Dates: Start 2024-01-21 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
endometrial thickness | day 12
  compare endometrial thickness among 3 group

SECONDARY OUTCOMES:
endometrial thickness difference between day 8 and day 12 | between day 8 and day 12
  compare endometrial thickness day 8 and day 12
clinical pregnancy rate | 12 weeks
  seen FHB at 12 weeks
chemical pregnancy rate | 2 weeks after transfer
  hcg > 25 u
miscarriage rate | up to 12 weeks
  abortion < 12 weeks
cancellation rate | day 14
  cancel cycle from thin endometrium < 7 mm

CONTACTS AND LOCATIONS:
Overall Officials: Sootthinan Pothisan, Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital, Bangkok Noi, Bangkok, Thailand